CLINICAL TRIAL: NCT01684670
Title: Intensive Dysarthria Sessions in Adults and Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Rhode Island (Other); University of Florida (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00039730
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Dysarthria; Down Syndrome
MeSH Terms: conditions — Dysarthria; Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral speech treatment (Experimental)
  Interventions: Behavioral: Speech sessions

INTERVENTIONS:
Behavioral: Speech sessions — Subjects will be instructed to use clear speech and increased effort when speaking.

SUMMARY:
This research study is designed to investigate the feasibility and treatment effects of a behavioral speech treatment in adults and children with Down Syndrome (DS) and dysarthria. The speech sessions will provide an intensive, articulation-based intervention focused on increasing effort during speech production via use of "clear speech." A single subject multiple baselines across subjects design will be employed in a total of six subjects divided into two groups of three. Changes in dependent measures will be determined by visual inspection, effect size determination, and time series analysis. The study follows accepted procedures in rehabilitation treatment and research and there are minimal foreseeable risks associated with participation.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children with Downs Syndrome and dysarthria
* Ages 8 years and older
* Ability to verbally communicate; follow simple commands and/or imitate others; hear speech at a conversational level; and participate in assessment and speech sessions activities

Exclusion Criteria:

* Additional serious medical problems which prevent meaningful participation in the study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility | 3-6 months
  Speech intelligibility in sentences scored by naive listeners.

CONTACTS AND LOCATIONS:
Overall Officials: Harrison N Jones, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States